CLINICAL TRIAL: NCT07206459
Title: Diaphragm Strength and Lung Volumes
Acronym: DIAVOLA
Status: Active, not recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 24-170
Record Dates: First submitted 2025-09-15; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-11

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Adults: Healthy participants will be recruited by work of mouth from the Grand Toronto Area.
  Inclusion criteria for the healthy participants will be age ≥18 years, no acute or chronic condition impacting respiratory, musculoskeletal or neurological system or that would interfere with the performance of the tests; body mass index <35 kg/m2 and sufficient English fluency to provide informed consent and to follow the study protocols.
  Exclusion criteria for the healthy participants will be contraindication for PNS (e.g., cardiac pacemaker or implanted defibrillator, cervical implants), contraindication for a nasogastric tube (e.g., esophageal varices, recent nasal bleeding)and pregnancy.
  Interventions: Other: Healthy Patients
- Critical Care Patients: Adult patients admitted to St. Michael's Hospital ICU, Unity Health Toronto, Ontario, Canada, Inclusion criteria for patients will be intubation for more than 6 hours, triggering or not the ventilator (any mode of ventilation).
  Exclusion criteria for patients will be primary contraindication for magnetic PNS, severe neurological disorders, pregnancy, current use of continuous neuromuscular blocking agents at the time of the study procedure, P/F ratio <120, unstable hemodynamics (2 vasopressors), monitored ICP.
  Interventions: Other: Critically Care Patients

INTERVENTIONS:
Other: Healthy Patients — RESEARCH DESIGN AND METHODS This will be a physiological observational study
  Study design. Participants will breathe on CPAP with a ventilator. The investigators will deliver the PNS at PEEP levels of zero cmH2O (baseline EELV), zero cmH2O + an abdominal binder (to reduce lung volume), five cmH2O and ten cmH2O. The abdominal binder will be used to achieve an EELV lower than at baseline. At the end of the protocol another PNS at zero cmH2O (baseline EELV) will be performed. Healthy participants will be exposed to the different levels of PEEP from 2 to 5 minutes before each PNS is performed.
  At every PEEP level, relative changes in EELV (∆z) will be measured with Electrical Impedance Tomography (EIT) to record relative changes in EELV and the electrical activity of the costal diaphragm will be measured using surface electromyography
  Groups: Healthy Adults
Other: Critically Care Patients — RESEARCH DESIGN AND METHODS This will be a physiological observational study
  Study design. For patients. The investigators will perform PNS at the patients own mode of ventilation at their clinical level of PEEP (baseline EELV), PEEP of zero cmH2O (if acceptable for 5 minutes), clinical PEEP ± 2 - 4 cmH2O. At the end of the protocol, another stimulation at the clinical level of PEEP (baseline EELV) will be performed. Patients will be exposed to the different levels of PEEP from 2 to 5 minutes before each PNS is performed.
  Groups: Critical Care Patients

SUMMARY:
Diaphragm dysfunction (loss of diaphragm strength) is common in the intensive care unit (ICU) patients using ventilators. The diaphragm is the main muscle of respiration and its dysfunction can prolong mechanical ventilation and increase mortality risk. The ventilator settings determine how much air and pressure the patient gets every breath and how much air is left on the lungs after they breathe out. The amount of air left on the lungs influence diaphragm strength measurements which can affect clinical decisions, such as weaning patients off ventilators. This research aims to explore the relationship between the amount of air left in the lungs and diaphragm strength to create a method of correcting measurements of diaphragm strength according to how much air the patients have in the lungs after they breath out. The investigators will test healthy individuals to understand this relationship, then verify if it holds true for ventilated patients by comparing results from both groups.

DETAILED DESCRIPTION:
Our ultimate objective is to create a correction factor for adjusting values of diaphragm strength obtained from measurements of pressure generated by PNS performed at various EELV induced by different levels of PEEP. This correction factor will be derived from the slope of the relationship between PEEP/EELV and diaphragm strength. The initial development of the correction factor will be conducted in healthy individuals, and its applicability will be assessed in mechanically ventilated patients. To achieve this, the investigators will compare the relationship between PEEP/EELV and diaphragm strength, measured through PNS, between both healthy subjects and individuals undergoing mechanical ventilation.

RESEARCH DESIGN AND METHODS This will be a physiological observational study

Study design. Healthy participants and patients will breathe on CPAP with a ventilator. The investigators will deliver the PNS at PEEP levels of zero cmH2O (baseline EELV), zero cmH2O + an abdominal binder (to reduce lung volume), five cmH2O and ten cmH2O. The abdominal binder will be used to achieve an EELV lower than at baseline. At the end of the protocol another PNS at zero cmH2O (baseline EELV) will be performed. Healthy participants will be exposed to the different levels of PEEP from 2 to 5 minutes before each PNS is performed.

At every PEEP level, relative changes in EELV (∆z) will be measured with Electrical Impedance Tomography (EIT) to record relative changes in EELV and the electrical activity of the costal diaphragm will be measured using surface electromyography . The (potentiated) PNS will be performed by bilateral anterior magnetic stimulation. Potentiation will be achieved by performing a maximum inspiratory pressure maneuver (MIP; healthy volunteers).

For patients. The investigators will perform PNS at the patients own mode of ventilation at their clinical level of PEEP (baseline EELV), PEEP of zero cmH2O (if acceptable for 5 minutes), clinical PEEP ± 2 - 4 cmH2O. At the end of the protocol, another stimulation at the clinical level of PEEP (baseline EELV) will be performed. Patients will be exposed to the different levels of PEEP from 2 to 5 minutes before each PNS is performed. At every PEEP level, relative changes in EELV (∆z) will be measured with Electrical Impedance Tomography (EIT) to record relative changes in EELV and the electrical activity of the costal diaphragm will be measured using surface electromyography . The PNS will be performed by bilateral anterior magnetic stimulation. Potentiation, when possible (patients triggering the ventilator), will be achieved by performing an end-expiratory occlusion maneuver on the ventilator for up to 30 sec or at least 3 inspiratory efforts.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the healthy participants will be age ≥18 years, no acute or chronic condition impacting respiratory, musculoskeletal or neurological system or that would interfere with the performance of the tests; body mass index <35 kg/m2 and sufficient English fluency to provide informed consent and to follow the study protocols.
* Inclusion criteria for patients will be intubation for more than 6 hours, triggering or not the ventilator (any mode of ventilation).

Exclusion Criteria:

* Exclusion criteria for the healthy participants will be contraindication for PNS (e.g., cardiac pacemaker or implanted defibrillator, cervical implants), contraindication for a nasogastric tube (e.g., esophageal varices, recent nasal bleeding)and pregnancy.
* Exclusion criteria for patients will be primary contraindication for magnetic PNS, severe neurological disorders, pregnancy, current use of continuous neuromuscular blocking agents at the time of the study procedure, P/F ratio <120, unstable hemodynamics (2 vasopressors), monitored ICP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 healthy adults and 15 critically ill adult patients admitted to St. Michael's Hospital ICU, Unity Health Toronto, Ontario, Canada. Healthy participants will be recruited by work of mouth from the Grand Toronto Area.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in diaphragm strength | Day 1 (within 5 minutes at each PEEP level during the intervention)
  Change in the pressure generated by the diaphragm (cmH₂O), assessed during end-expiratory occlusion on mechanical ventilation while applying phrenic nerve stimulation. Measurement will be obtained repeatedly on Day 1, between 3-5 minutes after each PEEP adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, PhD, Principal Investigator — Unity Health Toronto - St. Michael's Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due participant confidentiality.